CLINICAL TRIAL: NCT02303275
Title: Comprehensive 12-week Lifestyle Change Program in Elderly Patients With Heart Failure
Brief Title: Lifestyle Change Program in Elderly Patients With Heart Failure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Scripps Center for Integrative Medicine (Other)
Responsible Party: Principal Investigator, Eva Stuart, RN, Christopher Suhar, MD, Scripps Center for Integrative Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: LSCP_CHF_Suhar
Record Dates: First submitted 2014-11-20; First posted 2014-11-27 (Estimated); Last update posted 2014-11-27 (Estimated); Status verified 2014-11

CONDITIONS: Heart Failure
Keywords: Heart Failure; Congestive Heart Failure; Lifestyle Change
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lifestyle Change (Other): Lifestyle Change
  Interventions: Behavioral: Lifestyle Change

INTERVENTIONS:
Behavioral: Lifestyle Change — Intervention: Lifestyles Change Program (LCP)
  The LCP is a 12-week multi-disciplinary program that incorporates a holistic approach to chronic disease management, which will be tailored to our study population, patients with chronic heart failure. The core of the LCP includes:
  Clinician, Dietician, Exercise physiologist, Counselor, Nurse Case Manager Medical oversight by board-certified Cardiologist, Exercise prescription, Stress management classes (yoga, meditation, guided imagery), Group support, lifestyle change lectures, body composition analyses, grocery store tour, cooking classes, Music Wellness, and resiliency classes.
  Other Names: Integrative Medicine 12-week Lifestyle Change Program
Behavioral: Lifestyle Change — The lifestyle change program consists of classes conducted three times a week for 12 weeks at the Scripps Center for Integrative Medicine. Each day participants will spend about four to five hours in a variety of classes such as monitored exercise, group support, mindful-yoga and meditation, vegetarian cooking classes, music-centered wellness, mind-body lectures, and resiliency training.
  Other Names: Integrative Medicine Lifestyle Change Program

SUMMARY:
Summary

Chronic heart failure continues to be one of the highest economic burdens in the United States, heavily influenced by frequent readmissions to the hospital. This study will examine whether patients 65 years and older, who have NYHA class II and III heart failure, will improve their symptoms after participating in a comprehensive 12-week lifestyle change program. The investigators will recruit potential subjects primarily from the Scripps Clinic heart failure clinic at the Torrey Pines campus. Qualifying subjects will be randomized to medical treatment as usual or the lifestyle program. The investigators will enroll 17 subjects into each group which will provide 80% power and an alpha of 0.05.

The lifestyle change program consists of classes conducted three times a week for 12 weeks at the Scripps Center for Integrative Medicine. Each day participants will spend about four to five hours in a variety of classes such as monitored exercise, group support, mindful-yoga and meditation, vegetarian cooking classes, music-centered wellness, mind-body lectures, and resiliency training.

The primary outcomes will focus on determining functional status and physical agility using the 6-minute walk test, handgrip strength, and NYHA class categories. In addition, the investigators will capture subjective physical status with a self-reported questionnaire. Cognitive assessment will be performed using the Montreal Cognitive Assessment tool. To capture the subject's overall self-reported improvement the investigators will use a quality of life and a depression questionnaire. Secondary endpoints include hospital admission rates and all-cause mortality.

DETAILED DESCRIPTION:
The investigators Research Question and Hypothesis is as follows:

Comprehensive, evidence-based lifestyle and psychosocial interventions over a 12-week period (Lifestyles Change Program) can improve various objectives (6-minute walk distance, Left Ventricular Ejection Fraction (LVEF), New York Heart Association Class, grip strength, and cognitive function) as well as subjective (Quality of life, depression and functional screening) measures in patients with chronic heart failure. Secondary endpoints would include data such as hospital admission rates and all-cause mortality.

Background/ Gaps in Knowledge Chronic heart failure continues to be one of the highest economic burdens in the United States, heavily influenced by frequent readmissions. As a measure of performance quality, the Center of Medicare and Medicaid Services (CMS) began publically reporting hospital risk-standardized 30-day all-cause readmission rates, among fee-for-service beneficiaries discharged after hospitalization for heart failure from all the US acute care hospitals (1). Previous reported averages for hospital readmission in patients with chronic heart failure averages 25% to 30%, with some studies showing a readmission rate of up to 45% at 6 months.

There has been significant research examining various methods to reduce hospital admissions and improve functional capacity for patients with heart failure. Aside from published data on patient factors associated with readmission (age, sex, race, education, diabetes, renal disease, history of stroke, cognitive impairment, New York Heart Association (NYHA) class level, and serum markers [blood urea nitrogen, creatinine, C-reactive protein], etc), there have been many prospective studies evaluating readmission rates in CHF using interventions including: specialized multi-disciplinary teams (CHF nursing staff, pharmacists, physicians, etc), telephonic home monitoring, implantable device monitoring, various exercise programs (intermittent vs. continuous), meditation and spirituality, and early hospital follow-up.

Attempts at creating valid statistical models to predict patients at the highest risk for readmission used heterogeneous approaches and found substantial inconsistencies regarding which patient characteristics were predictive. From a policy perspective, as of 2009, a validated risk-standardized model to accurately profile hospitals using readmission rates is unavailable in the published English-language literature to date (3). Essentially, the identification of patients at high risk for heart failure readmission remains difficult with no validated objective assessment. Therefore, the strategy to reduce readmissions of heart failure patients is evolving to become a more personalized, patient-centered approach based on specific needs of each patient. For example, studies evaluating patient vs physician and healthcare staff perceptions for the causes of heart failure readmissions (using standardized questionnaires), shows discrepancy in the physician's opinion vs the patient's opinion about what factors influenced the readmission.

In essence, various aspects of the LCP have been evaluated in controlled clinical trials, but an overall, comprehensive study evaluating multiple components as included in the LCP has (to the investigators knowledge) not been done. Previous randomized controlled trials have shown benefit (6-minute walk, NYHA class, etc) using cardiac rehabilitation in patients with CHF (12). Yoga has been shown to improve exercise tolerance and positively affected levels of inflammatory markers in patients with CHF, with trends towards improvements in QoL (11). Education by a dietitian in patients with CHF has also been shown to result in a significant decrease in sodium intake compared with patients who simply receive written instructions (9). Studies have also evaluated spiritual well-being and depression in patients with heart failure, and have shown that greater spiritual well-being, particularly meaning/ peace was strongly associated with less depression (6). Interestingly, Tai Chi has been used in complimentary medicine for many years in patients with cardiovascular disease. Recently, a randomized study in 2011 showed that Tai Chi exercise improves quality of life, mood, and exercise self-efficacy in patients with CHF (5).

The investigators goal with the currently described study is to use a comprehensive, evidence-based Lifestyle Change Program (LCP) that incorporates all of the above individual components in a single program, individualized to each patient's physical abilities. Moreover, the investigators hypothesis is that such an intervention with chronic heart failure patients will improve Quality of Life, objective cardiometabolic markers, and reduce hospital admissions..

ELIGIBILITY:
Inclusions

1. Male or female, over 18
2. Able to commit to participating in the Lifestyle Change Program:

   * 4 -5 hours per day
   * 3 days per week
   * for a total of 12-weeks
3. History of CHF with systolic dysfunction (EF <45%) OR History of heart failure with preserved ejection fraction (HFpEF)
4. Must have had one previous admission for acute decompensated heart failure within the past year at time of enrollment.
5. New York Heart Association (NYHA) Class II - III symptoms:

   Class II: Mild symptoms (mild shortness of breath and/or angina) and slight limitation during ordinary activity.

   Class III: Marked limitation in activity due to symptoms, even during less-than- ordinary activity, e.g. walking short distances (20-100 m). Comfortable only at rest.
6. Labs: Complete Blood Count, Comprehensive Metabolic Panel must have been stable within the last 3 month.
7. Exercise: must be able to do some gentle exercises

Exclusions

1. Severe medical condition(s) that preclude participation in the Lifestyle Change Program
2. Unable to travel to the Scripps Center for Integrated Medicine Gym 3 times a week for 12 weeks
3. Severe cognitive, language, and psychosocial disabilities that prevent participation in the Lifestyle Change Program
4. Unsafe to participate in the exercise program based on the American College of Sports Medicine safety criteria such as:

   * Refractory chest pain
   * poorly controlled arrhythmias causing hemodynamic symptoms
   * high degree Atrioventricular block
   * pacemakers which do not permit adequate heart rate response to exercise
   * significant uncorrected primary vascular disease
   * isolated pulmonary hypertension
   * poorly controlled symptomatic postural hypotension
   * obstructive cardiomyopathies
5. Severe untreated anemia.
6. Participation in another research study in the last month
7. Smoking

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2013-05; Primary Completion 2016-05 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
Functional status as measured by the 6-minute walk test. | After 12-weeks
  Subjects randomized to the intervention group will receive a 12-week Lifestyle Change program intervention
Functional status as measured by handgrip strength. | After 12-weeks
  Subjects randomized to the intervention group will receive a 12-week Lifestyle Change program intervention
Functional status as measured by New York Heart Association class categories. | After 12-weeks
  Subjects randomized to the intervention group will receive a 12-week Lifestyle Change program intervention

SECONDARY OUTCOMES:
Hospital Admission Rates | During the intervention period of 12 weeks and for 1 year after completing the program.
  Secondary endpoints include hospital admission rates.
all-cause mortality | for 1 year after completing the intervention
  Secondary endpoints include all-cause mortality

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Suhar, MD, Principal Investigator — Scripps Center for Integrative Medicine; James Gray, MD, Study Director — Scripps Center for Integrative Medicine; James Heywood, MD, Study Chair — Scripps CHF Clinic, Torrey Pines Campus
Locations (1):
- Scripps Center for Integrative Medicine, La Jolla, California, United States